#### Walter Reed Army Institute of Research

#### CONSENT TO PARTICIPATE IN RESEARCH

Title of Protocol: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to

Evaluate the Safety, Tolerability, and Immunogenicity of Ranging Doses of SARS-CoV-2-Spike-Ferritin-Nanoparticle (SpFN\_1B-06-PL) Vaccine with Army Liposomal Formulation QS21 (ALFQ) for Prevention of

COVID-19 in Healthy Adults

**Sponsor:** U.S. Surgeon General, Department of the Army

**Principal** 

**Investigator:** Brittany Ober-Shepherd, M.D.

#### Introduction

Thank you for your interest in this research study. This study will take place at the Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center (CTC). This study is sponsored and funded by the United States Department of Defense. The box below provides important information about the study that you should think about before deciding to join the study. We will provide more detailed information below the box. Please ask questions about any of the information before you decide whether to participate. You may also wish to talk to others (for example, your family, friends, or your doctor) about this study, before agreeing to join. If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.

| Key Information | |
|---|---|
| Voluntary<br>Participation | You do not have to take part in this research. It is your choice. You may decide not to participate in the study, or you may decide to stop participating in the study at any time without penalty or loss of benefits to which you are entitled. |
| Purpose | We are doing this research to test an experimental vaccine for SARS-CoV-2, the virus that causes COVID-19 disease, because a safe and effective vaccine is needed to prevent this disease. We need to learn if the vaccine is safe and if it produces an appropriate immune response. Immune responses occur when your body recognizes and defends itself against foreign substances such as bacteria and viruses by making proteins that get rid of the foreign substances. These proteins are called antibodies. Vaccines also cause immune responses, but they help teach your body how to defend itself from a virus without infecting you with the virus. |
| Experimental<br>Products | There are 3 different products used in this study: 1. SpFN_1B-06-PL – the experimental vaccine against SARS-CoV-2, which has been tested in animals, but not yet in humans. |

| D. C | <ol> <li>ALFQ – the experimental adjuvant (explained later) that is added to the vaccine that has been used in humans but is still being tested.</li> <li>Normal saline (sterile salt water) will be the placebo (more on this later).</li> </ol> |
|---|---|
| Duration | You will be in this study for about 18 months or 1.5 years. |
| Procedures | If you participate in the study, you will: Be randomly assigned to get either the experimental COVID-19 vaccine or a placebo Receive 2 or 3 vaccine or placebo injections in the same arm muscle Group 1 and 2 will receive the injections on Study Days 1 and 29 (4 weeks) You will be notified by phone or by mail of your random assignment to either vaccine or placebo after the last active participant completes their Study Day 57 visit If you received vaccine on Study Days 1 and 29 and have not received a licensed COVID-19 vaccine or one given Emergency Use Authorization, you will be offered an optional third vaccination at Study Day 181 (6 months) If you are eligible, you can either agree to or decline receipt of the third vaccination at Study Day 181 Regardless of your decision and eligibility, you can continue to participate in all subsequent scheduled visits after Study Day 57 If you received placebo on Study Days 1 and 29, you are not eligible to receive an injection on Study Day 181 but can continue to participate in all scheduled visits after Study Day 57 Record any side effects that you may experience for 7 days after you receive the injections Record any side effects that you may experience for 7 days after you receive the injections Have blood, nose swabs, and saliva samples collected at each visit Have urine samples collected for pregnancy testing (females only) Undergo medical and physical examinations Answer questions about potential exposures to COVID-19 in your daily life |
| Risks | In this study, there may be risks associated with the vaccine, blood draws, and nose swabs. This vaccine has never been tested in humans, so not all risks are currently known. The most serious known risk is the possibility of a potentially lifethreatening allergic or (rare) autoimmune reaction to the vaccine. An autoimmune reaction occurs when your immune system malfunctions and produces antibodies that attack normal body tissues. You will be referred for care and treatment if you should develop an autoimmune reaction. The clinic has emergency medical equipment in place to handle both minor and potentially life-threatening allergic reactions if they should occur. There is also a theoretical concern that coronavirus vaccines might make |
| | COVID-19 disease worse. This theoretical concern is based on animal |

studies of 'inactivated vaccine' (a vaccine that contains a live, lab-grown virus that is not capable of causing an infection) for other coronaviruses such as SARS and MERS. This reaction was not seen in humans who received these vaccines. In addition, the vaccine in this study is not an inactivated vaccine; therefore, the possibility that a COVID-19 infection could be worsened after receiving the experimental vaccination should be very minimal. Since the experimental vaccine does not contain the virus, it cannot cause you to become infected with COVID-19.

There is no guarantee that you will be protected from COVID-19 infection from receiving the experimental vaccine and there is the possibility that you could receive the placebo, so you should continue to practice all exposure prevention measures including wearing a mask, practicing social distancing, and frequent hand washing. If you are informed that you received the placebo during this study, we encourage you to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization as soon as possible.

#### **Benefits**

This study is experimental, and there is no guarantee that you will receive any benefit from participating. As part of the study procedures, you will be tested for SARS-CoV-2 and undergo general health screenings, and some participants may benefit from knowing if the results of these tests indicate an infection or are abnormal.

#### **Alternatives**

The alternatives to participating in this study are to receive a licensed COVID-19 vaccine or one given Emergency Use Authorization, or participate in another study. At each visit, you will be asked if you have received any experimental COVID-19 vaccines outside of this study, licensed COVID-19 vaccines, or vaccines given Emergency Use Authorization. You will not be prevented or discouraged from receiving a licensed COVID-19 vaccine or one given Emergency Use Authorization, but to be eligible for participation in this study you must agree to not join another study that involves exposure to investigational or noninvestigational vaccines or products while in this study. If you choose to receive a licensed COVID-19 vaccine or one given Emergency Use Authorization prior to the last active participant completing Study Day 57, you can request that the study team inform you about whether you received the experimental vaccine or placebo. You will otherwise be notified about whether you received the experimental vaccine or placebo after the last active participant completes the Study Day 57 visit, and you may be offered an optional third vaccination if you are still eligible for the study. All participants will continue to be followed for safety purposes. If you are informed that you received placebo during the study or if you choose not to receive the optional third vaccination, you are encouraged to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization. If you choose to receive the optional third vaccination, you are still encouraged to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization, but you

| | should wait until at least 28 days have passed since the last injection. |
|---|---|
| Compensation | You will receive payment for your participation in this study. You will not receive compensation for missed or incomplete visits. |

## Why is this research being done?

We are doing this research to test an experimental vaccine to prevent infection with severe acute respiratory syndrome coronavirus (SARS-CoV-2), which causes the COVID-19 disease. SARS-CoV-2 is a new virus that is spreading from person-to-person throughout the world. COVID-19 symptoms can range from mild (or no symptoms) to severe illness. A safe and effective vaccine is needed to prevent disease and death from SARS-CoV-2 infection.

The experimental vaccine in this study contains 2 parts: the vaccine (called SpFN\_1B-06-PL) and an experimental adjuvant called ALFQ. An adjuvant is a substance added to vaccines that can help to make the vaccine more effective by improving the immune response or causing the immune response to last longer. We need to learn if this vaccine and the adjuvant combination is safe and produces an immune response that can teach your body to protect itself from COVID-19. The SpFN\_1B-06-PL part of the vaccine has been tested in animals; however, this will be the first time that it will be tested in humans. The ALFQ adjuvant has been tested in humans and has caused only minor or moderate side effects.

The experimental vaccine does not contain the virus and cannot cause you to become infected with the COVID-19 disease. The experimental vaccine has not been approved or cleared by the FDA; however, they have allowed its use in this research study to learn more about its safety and efficacy.

#### Who can participate in this study?

You may take part in this study if you are a healthy male or female between ages 18 and 55 years, not pregnant or breastfeeding, with a body mass index (a ratio based on your height and weight) between 18.1 kg/m<sup>2</sup> and 35.0 kg/m<sup>2</sup> who is willing and able to sign and date this informed consent form, can demonstrate an understanding of the study by achieving a passing score on a test of understanding within 3 attempts, is willing to comply with the study requirements, is available for the duration of the study, and is willing to provide a phone number at which you can reliably be contacted. Study staff will use your phone number to follow-up with you after you receive the vaccine or placebo injection, to remind you of upcoming study visits, and to reschedule any missed visits. We would also like to collect information for an emergency contact person that would be able to help us get in contact with you if we are unable to for any reason. Study staff will only use your emergency contact if we are unable to get in touch with you within 7 days after a missed visit as we want to make sure that you are safe. You must also be free of any significant medical problems, agree to not donate blood or plasma outside of this study for the duration of your participation in this study, and agree to the future use of your specimens. Female participants are required to undergo pregnancy testing, to not be pregnant, to not be breastfeeding, and to use an acceptable method of contraception from 30 days before enrollment until at least 60 days after the last injection (about 9 months in total) if of childbearing potential.

After signing the consent form to take part of the study, you will be asked to take a test of understanding to see how much you understand the study. You must answer at least 9 out of 10 questions correctly in order to participate in the study. You may take the test 3 times to get a score

of 9 out of 10. The doctor will then ask you questions and do a physical examination to see if there is any reason you should not join in the study.

You **cannot** join this study if you have:

- Current or prior COVID-19/SARS-CoV-2 infection
- HIV, hepatitis C, or hepatitis B infection
- An autoimmune disease or deficiency
- A history of organ and stem cell transplantation
- A history of cancer
- Diabetes (type I or II) and/or thyroid disease
- A chronic disease or condition including but not limited to asthma, autoimmune disease, sickle cell anemia, chronic hepatitis or cirrhosis, chronic pulmonary disease, chronic renal disease, and chronic cardiac disease including hypertension even if medically controlled
- A history of a serious allergic reaction to any vaccines, vaccine component, or latex
- A major surgery within a month before screening or plans to have a major surgery during the study
- Have a fever or illness within 48 hours before you are scheduled to receive a study injection, however you can be reassessed by a study doctor if your illness resolves within 7 days.
- Tattoos, scars, or other marks that would, in the opinion of the investigator's, interfere with the assessment of the vaccination site
- Received or plan to receive any of the following:
  - o Blood products within 3 months prior to enrollment or at any time during the study
  - An experimental COVID-19 vaccine outside of this study, a licensed COVID-19 vaccine or a COVID-19 vaccine that has been given Emergency Use Authorization from the FDA
  - Any "live-attenuated" vaccine (e.g., oral polio, yellow fever, measles, etc.) within 30 days prior to enrollment in the present study or until 30 days after the last vaccination
  - Any killed or inactivated vaccine (e.g., injected polio, hepatitis A, rabies, pertussis, etc.) within 14 days prior to enrollment in the present study or until 30 days after the last vaccination
    - Note: You are allowed to get a flu shot during your participation in this study as long as it is given at least 14 days prior or 30 days after each study injection
  - Experimental research drugs from another study within 3 months prior to enrollment in the present study or at any time during your participation in this study.

In addition to the above, you may not participate in the study if you are emergency medical services personnel or a healthcare provider who has contact with patients in a potentially high risk/high exposure setting, currently smoke cigarettes and/or vape, or if you have a history of any condition(s) that, in the opinion of the investigators, may interfere with your full participation in the study or that may impair your ability to provide informed consent.

Volunteers who are active duty military personnel must receive written approval from their supervisor prior to participating in the study, per WRAIR Policy Letter 12-28. For volunteers who are DoD-affiliated, an ombudsperson will be present when recruitment is done in a group setting.

The ombudsperson acts as an impartial and objective advocate for individuals participating in research.

## How many people will be in the study?

This study was initially designed to have a total of 72 people take part in this study. If 72 people enrolled, 60 would receive the experimental COVID-19 vaccine and 12 would receive a placebo. At this time, no more people will be enrolled in the study, but follow-up visits will continue for safety purposes.

### How long will I be in the study?

About 18 months (1.5 years)

### What will happen during this study?

If you are selected to participate in the study, you will be randomly assigned (by chance) to get either the experimental COVID-19 vaccine or a placebo. The placebo is a sterile saltwater injection that contains no vaccine intended to prevent COVID-19. Neither you nor the study doctor and staff will know whether you have received the experimental COVID-19 vaccine or placebo until after the last active participant completes the Study Day 57 visit. Once that happens, you will be notified by phone or mail about whether you received the experimental vaccine or placebo and if you received the experimental vaccine, which dose you were given. You can request this information earlier if you choose to receive a licensed COVID-19 vaccine or one given Emergency Use Authorization, but you will not be able to receive any further study injections after receiving a licensed COVID-19 vaccine or one given Emergency Use Authorization.

If you are eligible and choose to participate in this study, you will be enrolled into one of the following study groups:

- **Group 1:** 25 μg SpFN\_1B-06-PL + 0.5 mL ALFQ (20 participants) or Placebo (4 participants) in a total 1.0 mL injection volume at Study Days 1 and 29. Optional 25 μg SpFN\_1B-06-PL + 0.5 mL ALFQ (20 participants) at Study Day 181 for participants who received the investigational vaccine at Study Days 1 and 29.
- Group 2: 50 μg SpFN\_1B-06-PL + 0.5 mL ALFQ (20 participants) or Placebo (4 participants) in a total 1.0 mL injection volume at Study Days 1, 29, and 181. Optional 50 μg SpFN\_1B-06-PL + 0.5 mL ALFQ (20 participants) at Study Day 181 for participants who received the investigational vaccine at Study Days 1 and 29.

Enrollment will go slowly, in a stepwise approach so that we can closely monitor any safety concerns during regular health reviews. These steps are detailed in the table below.

| Step 1 Group 1 | 3 people will get the 25 μg dose of the vaccine 1 person will get the Placebo | Four participants will receive the study injection and be followed closely for symptoms or reactions for seven days. |
|---|---|---|
| Step 2<br>Group 1 | <ul><li>17 people will get the 25 μg dose of the vaccine</li><li>3 people will get the Placebo</li></ul> | If there are no safety concerns after the seven-day review in <b>Step 1</b> , 20 more participants will receive the study injection and be followed closely for |

| | | symptoms or reactions for seven days. |
|---|---|---|
| Step 3 Group 2 | 3 people will get the 50 μg dose of the vaccine 1 person will get the Placebo | If there are no safety concerns after the seven-day review in <b>Step 2</b> , four participants will receive the study injection and be followed closely for symptoms or reactions for seven days. |
| Step 4 Group 2 | <ul><li>17 people will get the 50 μg dose of the vaccine</li><li>3 people will get the Placebo</li></ul> | If there are no safety concerns after the seven-day review in <b>Step 3</b> , up to 20 more participants will receive the study injection and be followed closely for symptoms or reactions for seven days. |

### If you agree to take part in this research, you need to agree to the following:

There are at least 12 required clinic visits and up to 5 scheduled phone or video (if your phone or computer have video capability) visits over approximately 18 months. The scheduled phone or video visits will be completed in the days following each study injection so that the study team can both collect information about any side effects that you may have experienced as well as to ensure your safety. In addition to the scheduled clinic and phone or video visits, you may be asked to come in for additional visits if you develop symptoms that are concerning to you or the study team, or repeat testing is needed. Transportation to and from the in-person clinic visits via a car or van service is available for all participants within 250 miles of the clinic. This transportation will be coordinated and paid for by the study team and will not affect the compensation that you receive for participating. If you would like to use this service, please tell a member of the study team.

Over the first 6 months, you will receive 2 or 3 injections into the same muscle of your arm. If you receive the investigational vaccine at Study Days 1 and 29, you may be eligible to receive an optional third vaccine injection at Study Day 181. At each visit, you will provide blood, saliva, and nose swab samples. The amount of blood drawn at clinic visits will vary from about 2 tablespoons (29 mL) to about 5 tablespoons (71.5 mL), depending on the visit. You might also be asked to have laboratory tests completed between regular visits if needed to check your health. The total amount of blood drawn during the study will be about 3 cups (720.5mL to 763.5mL). Female participants will give a urine sample to check for pregnancy before each study injection. The Vaccine/Placebo Injection visits will take about 2-3 hours, follow-up visits will take up to an hour, and telephonic follow-up visits will take about 5 minutes.

## What are my responsibilities during the study?

If you participate in this study, you will be asked to:

- Sign the informed consent form and achieve a passable score (9 out of 10 correct) on the Test of Understanding.
- Provide complete and accurate information about any current or past medical conditions, medications you have been taking or are taking now. For your safety, you must inform study staff of any new medical conditions or medications that begin during your participation in the study.

- Attend all scheduled visits and follow all of the study doctor's instructions.
- Be available for telephone calls from the study staff. If you cannot keep an appointment, contact the study clinic immediately to reschedule.
- Provide contact information for someone who might be able to help us get in contact with you if we are unable to get in touch with you for any reason.
- Quickly inform the study doctor or study staff of any health problems, even if you think the vaccine did not cause them.
- Have blood, saliva, and nose swab samples taken at every visit.
- Complete the diary card daily, as instructed by the study doctor and staff. You will get a ruler to measure any injection site reactions. Bring the diary card to each visit.
  - We may ask to photograph a visible reaction and that you take part in a video follow-up visit if you have that capability on your phone or computer.
- Take and record your body temperature in the diary card daily during the seven days after each injection with the thermometer provided. If you feel ill after Day 8, you need to continue to record any symptoms.
- Not enroll in ANY other clinical research study in which you would receive an investigational or non-investigational vaccine/product while you are in this study.

You will be given a study schedule that contains details about what will happen at each visit. The procedures and tests described in the schedule are part of the study; therefore, if you do not agree to these procedures and tests, you cannot participate in this study.

#### What precautions do I need to take?

There several precautions that you need to take during this study to reduce possible risks and to ensure that the scientific study results are accurate.

- Female participants must not be pregnant or breastfeeding and, if of childbearing potential, must have used an effective form of contraception for at least one month before starting this study. This contraceptive method must be used until at least two months after the last study injection. Acceptable contraceptive methods for female participants include:
  - o Hormonal contraceptives (such as pills, injections, patches, implants, and others) that inhibit ovulation
  - o Intrauterine device
  - o Intrauterine hormone-releasing system
  - o Prior bilateral tubal occlusion
  - o A male partner who has previously undergone a vasectomy
  - o Abstinence from penile-vaginal intercourse
- All participants should continue to practice all exposure prevention measures including
  wearing a mask, practicing social distancing, and frequent hand washing. Participants who
  become infected with COVID-19 during the study will not be eligible to receive further
  study injections.

## What will happen to my samples during this study?

**Blood, saliva, nose swabs, and urine specimens:** The investigators will obtain blood, saliva, and nasal swabs to test for any possible side effects as well as evaluate the immune response to the vaccine. Nasal swabs collected in this study will be used to test for COVID-19 infection. Urine collected at study visits will be used for pregnancy tests for female volunteers.

**HLA and genetic tests:** Part of the blood samples for this study will be used to analyze for HLA ('Human Leukocyte Antigen') type. HLA is a group of proteins present on the surface of all cells in the human body with an important role in the immune response to infection. Determining HLA type is necessary to be able to perform certain research studies. We will not notify you with the results of this test. The HLA test for this study is not a normal medical test and the test result cannot be used for treatment purpose.

## What will happen to my samples after this study?

During your participation in this study, blood, saliva, and nose swab samples will be collected from you as already explained. We will store left over samples in a secure central storage site (not in the clinic) for future research to learn more about SARS-CoV-2 and COVID-19, vaccines, the immune system, and/or other medical conditions. Future research on your samples may include genetic testing. There are no plans to notify you of the results of future genetic testing as the testing will be done only for research purposes and the tests that will be used are not approved for use in making health care decisions.

Specimens will be stored and labeled with a numeric barcode without your name or other personally identifiable information attached. Only authorized personnel are able to connect those numeric codes and your name. Personally Identifiable Information will be kept confidentially according to all applicable laws and regulations.

Your samples may also be sent to collaborators outside of WRAIR and/or internationally. Your personal information will not be sent to collaborators, so they will not be able to identify you as an individual. Your samples may be used for future research studies or distributed to another investigator for future research studies without obtaining additional informed consent from you. If required by law or policy, future research that uses stored samples must be reviewed and approved by an Institutional Review Board (IRB), which is a committee that is responsible for overseeing the safety, welfare, and rights of research participants.

Your samples will not be sold or used directly to develop any commercial product. The results of this study could play a role in whether the FDA will approve the vaccine for sale at some time in the future. You will not receive money or other compensation should this occur.

#### What are the possible risks and discomforts?

This section describes the risks associated with the experimental SARS-CoV-2 vaccine and other study procedures. There may be additional risks related to the experimental SARS-CoV-2 vaccine that are currently unknown. If we learn about new risks during this study, we will tell you.

**Possible** risks from the injection: Temporary stinging, pain/tenderness, hardness, redness, soreness, itchiness, swelling or bruising at the injection site on your arm. There is a very small chance of infection.

**Possible** risks from any vaccine: Fever, chills, rash, aches and pains, nausea, headache, and fatigue. These types of reactions are usually greatest within the first 24 hours after vaccination and may last 1 to 3 days. While rare, there is also the possibility of a serious, even life-threatening, allergic reaction as may occur with the administration of any vaccine. The clinic has emergency medical equipment available to handle both minor and potentially life-threatening allergic reactions.

**Possible** risks of the experimental SARS-CoV-2 vaccine: The risks of the experimental vaccine are unknown, however in addition to the above there is a possibility you may experience diarrhea, difficulty breathing, cough, nasal drainage, nasal congestion, or a sore throat.

Experimental vaccines or adjuvants could uncover or worsen an immune-related disease or syndrome and there is a theoretical concern that coronavirus vaccines might make COVID-19 disease worse. This theoretical concern is based on animal studies of 'inactivated vaccine' for other coronaviruses such as SARS and MERS. This reaction was not seen in humans who received these vaccines. In addition, the vaccine in this study is not an inactivated vaccine; therefore, the possibility that a COVID-19 infection could be worsened after receiving the experimental vaccination should be very minimal.

While rare, there is also the possibility that you may develop inflammation of the heart muscle or inflammation of the lining outside the heart. Most of the cases of this inflammation after vaccination have been in males under 40 years old after the second dose of an mRNA vaccine, but cases have also been reported in older males, in females, and following other doses. Symptoms of this inflammation typically appear within a week of receiving the vaccine but may be experienced up to 6 weeks after vaccination and include chest pain, shortness of breath, or feelings of having a fast-beating, fluttering, or pounding heart. If you experience any of these symptoms, please seek immediate medical attention and inform the study team when possible. This risk is based on reported side effects from mRNA COVID-19 vaccines. The vaccine in this study is not an mRNA vaccine, therefore this risk is very minimal.

*Unknown* safety risks: This vaccine has never been tested in humans so there may be unknown side effects – even serious or life-threatening risks – that we do not yet know about. Please tell the study staff as soon as possible about any side effect you think you are having that may be serious or cause concern. This is important for your safety.

It is currently unknown if the experimental vaccination will protect you from COVID-19 infection and there is the possibility that you could receive the placebo, so you should continue to practice all exposure prevention measures including wearing a mask, practicing social distancing, and frequent hand washing. If you are informed that you received the placebo during this study, we encourage you to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization as soon as possible.

**Possible** risks of blood draws: Pain, bleeding, bruising, feeling lightheaded, fainting, or rarely, infection at the site where the blood is taken. To minimize the risks, trained health care providers will draw your blood.

**Possible** risks to Pregnancy: If you are pregnant or breast-feeding, then you cannot participate. We do not know the possible effects of the study vaccine on the unborn baby or nursing infant. Therefore, female participants must have a negative pregnancy test before the study vaccination and, if of childbearing potential, agree to use contraception beginning at least 30 days prior to

receiving the first study injection until at least 60 days after the last injection. You must notify the clinic staff immediately upon learning that you have become pregnant during this study. You must also notify the clinic if you suspect that you **might** be pregnant during this study. You will be asked to continue with the planned study follow-up visits for safety purposes and contacted later to learn about the outcome of any pregnancy that starts in the first 60 days after a study vaccination.

**Possible** risks from nose swabbing: Nose swabbing may cause discomfort and sometimes can cause your nose to bleed. This discomfort is minimized by having a trained nurse or physician perform these collections for you.

**Possible** risks from genetic testing: The greatest risk associated with genetic testing is your privacy. Genetic test results can be used to provide information about how susceptible you are to certain diseases. Used inappropriately, this information could be discriminatory (for example, by insurance companies). HLA typing can also be used to figure out who the true parent of a child is (if compared to the child's HLA type). However, the risk of this happening is extremely low, because your results will not be part of your medical records and will only be labeled with your study number rather than any of your personal information. Neither you nor your doctor will get the results as the tests are for research purposes only and not used to make health-related decisions.

In this study, we will not look at your full set of genes; we would assess specific genes that vary from person to person related to immune responses after vaccination.

You should know that Federal law, called the Genetic Information Nondiscrimination Act (GINA), generally prohibits health insurance and employment discrimination based on your genetic information. Health insurance companies and group health plans may not use your genetic information when making decisions about your eligibility or premiums. GINA's health insurance protections do not apply to members of the military who receive their healthcare through Tricare, to veterans who receive their healthcare through the Veterans' Administration, or to Federal employees who get their care through Federal Employee Health Benefit Plans. However, these groups may have policies in place that provide similar protections.

Employers with 15 or more employees may not use your genetic information when deciding to hire, promote, or fire you or when setting the terms of your employment. While GINA's employment protections do not apply to military members and Federal employees, presently, an Executive Order protects federal employees from genetic discrimination in employment, and the military has its own policies in place that may protect against genetic discrimination.

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

Once information that personally identifies you is removed from your data or specimens, then your data or biological samples may be used for future research studies or given to other researchers for future research studies without your permission to do so. If you stop taking part, the data and samples collected during your participation will continue to be used.

*Other* Risks: You may not donate blood outside of this study for the duration of your participation in this research study.

#### What are the possible benefits from being in this research?

This study is experimental, and there is no guarantee that you will get any benefit from it. As part of the study procedures, you will be tested for SARS-CoV-2 and undergo general health screenings, and some participants may benefit from knowing if the results of these tests indicate an infection or are abnormal. As noted in the next section, we will alert you if you test positive for COVID-19, HIV, or hepatitis; otherwise, we will only share results with you if specific test results are abnormal.

### What if new information is learned about my health?

As part of the research study, we will take blood samples to check your general health. We will share any abnormal test results with you as long as the tests are approved for clinical decision-making and the results indicate that medical intervention may be necessary. You may have a copy of these lab results if you wish. You will regularly be tested for COVID-19 while you are in this study and positive results must be reported to the Maryland Department of Health. If you test positive for COVID-19 during the study, you will be alerted of the result but you will not be able to receive any further study injections. Even though you won't receive any further study injections, we request that you continue to attend study visits so that the study staff can monitor your health for safety purposes. This follow-up will be done only if you are willing and if you are healthy so as not to expose others to COVID-19. If the study staff determine that in-person visits are unsafe, then a portion of these follow-up visits can be completed by phone and/or video. Any positive HIV and hepatitis results must also be reported to the Maryland Department of Health; however, you will only be tested for those at the screening visit. You will also be alerted if you test positive for HIV or hepatitis.

## What are my other options if I do not take part in this study?

The alternatives to participating in this study are to receive a licensed COVID-19 vaccine or one given Emergency Use Authorization or participate in another study. At each visit, you will be asked if you have received any experimental COVID-19 vaccines outside of this study, licensed COVID-19 vaccines, or vaccines given Emergency Use Authorization. You will not be prevented or discouraged from receiving a licensed COVID-19 vaccine or one given Emergency Use Authorization, but to be eligible for participation in this study, you must agree to not join another study that involves exposure to investigational or non-investigational vaccines or products while in this study. If you choose to receive a licensed COVID-19 vaccine or one given Emergency Use Authorization prior to the last active participant completing Study Day 57, you can ask the study team to inform you about whether you received the experimental vaccine or placebo. You will otherwise be notified about whether you received the experimental vaccine or placebo after the last active participant completes the Study Day 57 visit, and you may be offered an optional third vaccination if you are still eligible for the study. All participants will continue to be followed for safety purposes. If you are informed that you received placebo during the study or if you choose not to receive the optional third vaccination, you are encouraged to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization. If you choose to receive the optional third vaccination, you are still encouraged to get vaccinated with a licensed COVID-19 vaccine or one given Emergency Use Authorization, but you should wait until at least 28 days have passed since the last injection.

## Will I have to pay for anything if I take part in this research?

You will not be responsible for any of the costs associated with the study procedures, however you

will have to pay for your transportation to and from the clinic if you don't use the study-provided transportation. You will also need to have access to a phone.

## Will I be paid to take part in this research?

You will be compensated for your time and effort as follows:

- \$200 screening visit
- \$250 vaccine/placebo injection visit (participants who do not receive the optional third injection for any reason will still receive \$250 for completing the Study Day 181 visit)
- \$150 for each follow-up visit (including unscheduled clinic visits)
- \$25 Phone/video visit
- \$200 bonus for completing the study

The total compensation that you can receive for participating in this study, if there are no missed or incomplete visits, is \$2475. Transportation to and from the in-person clinic visits via car or van service will not affect the compensation amounts listed above. You will not receive compensation for missed or incomplete visits.

In addition to the amounts listed above, you will be compensated \$150 for unscheduled visits that may be requested by the study investigator, that may be required to repeat lab tests to verify/clarify results or to better evaluate abnormal lab values, to evaluate a research-related injury or illness, or to collect specimens that could not be collected at a scheduled study visit.

By regulation, active duty personnel and federal employees who are on duty can be compensated only for visits in which blood draws occur, at a rate of \$50 per visit. Active duty personnel and federal employees who are off duty or on leave may be compensated at the same rate as other study participants.

You can earn additional compensation for directing others who may be interested in this study to contact the CTC. You will receive \$75 for each referred person who then attends a screening session and meets all inclusion and none of the exclusion criteria. This compensation is independent of the referred person's decision to enroll.

Other than medical care that may be provided and other payment specifically stated in this form, there is no other compensation available for you taking part in this study.

## What happens if I am injured because of taking part in this research?

If, at any time, you believe you have suffered an injury or illness because of taking part in this research, please contact the PI, Dr. Brittany Ober-Shepherd, at 260-438-9948 or 301-500-3636.

If you are injured because of your participation in this research and you are a DoD healthcare beneficiary (e.g., active duty military, military spouse, dependent of active duty military, retiree), you are entitled to medical care for your injury within the DoD healthcare system, as long as you remain a DoD healthcare beneficiary. This care includes but is not limited to free medical care at DoD hospitals or clinics.

If you are injured because your participation in this research, and you are not a DoD healthcare beneficiary, you are entitled to care for your injury at an Army hospital or clinic; medical care charges for care at an Army hospital or clinic will be waived for your research-related injury. You

are also entitled to care for your injury at other DoD (non-Army) hospitals, but such care for your injury at other DoD (non-Army) hospitals or clinics may be time-limited, and your insurance may be billed. It cannot be determined in advance in which Army or DoD hospital or clinic will provide care. If you obtain care for research-related injuries outside of an Army or DoD hospital or clinic, you or your insurance are responsible for medical expenses.

For DoD healthcare beneficiaries and non-DoD healthcare beneficiaries: Transportation to and from hospitals or clinics will not be provided, except in emergencies or if a non-DoD healthcare beneficiary requires a military escort for access to the DoD medical facility.

Due to the COVID-19 public health emergency, the federal government has issued an order that may limit your right to sue if you are injured or harmed while participating in this COVID-19 study. This order limits your right to sue researchers, healthcare providers, any study sponsor, manufacturer, distributor or any other official involved with the study. However, the federal government has a program that may provide compensation to you or your family if you experience serious physical injuries or death. To find out more about this "Countermeasures Injury Compensation Program" please go to https://www.hrsa.gov/cicp/about/index.html or call 1-855-266-2427.

Other than any compensation that you may receive from the "Countermeasures Injury Compensation Program", there is no additional compensation available for research-related injuries or any medical expenses incurred for the treatment of research-related injuries.

If you believe you have had a research-related injury, please contact the PI. If you have any questions, please contact the PI. In addition, an emergency contact card will be provided to you with numbers to contact at any time.

# How will you protect my privacy and the confidentiality of records about me? We will take measures to protect your privacy, but we can never fully guarantee the protection of your privacy. We will try our best to protect your privacy by doing the following:

Your name and any identifiable information (for example, your address or social security number) will not be part of the study data. Your biological samples are labeled only with an identification code that consists of numbers and letters. Only the study investigators, study coordinators, and representatives from certain agencies (listed below) will be allowed to know which codes belong to you and to have access to your study information. Your research chart, where your personal information is stored, will be kept secure, in a locked cabinet, inside a locked room, with limited access. This is the same with your electronic information or data stored on a computer – only a few authorized staff members have access to the password-protected, secure database.

Authorized representatives of the following groups may need to review your research and or medical records as part of their responsibilities to protect research participants:

- Walter Reed Army Institute of Research Institutional Review Board (IRB) responsible for review and oversight of human research
- The Department of Defense (DoD) and other Federal offices charged with regulatory oversight of human research
- Food and Drug Administration (FDA)

• U.S. Army Medical Research and Development Command (USAMRDC)

For volunteers in the military, information bearing on your health may need to be reported to appropriate medical or command authorities. For example, if you share with us that you are feeling suicidal or homicidal, we may need to report this.

Research and clinical information relating to you will be shared with other investigators and the scientific community through presentation or publication; however, you will not be identified by name or other personal information that could be used to identify you.

#### **Clinical Trial Information**

A description of this clinical trial will be available on http://www.ClinicalTrials.gov as required by U.S. Law. This website will not include information that can be used to identify you. At most, the website will include a summary of results. You can search this website at any time.

## What if I decide not to take part in this research?

It is your choice whether or not you want to take part in this research.

If you decide to take part, you can stop taking part in this research at any time without any penalty or loss of benefits to which you are entitled. Deciding not to take part now or withdrawing later does not harm, or in any way affect, your medical care or future relationship with the Walter Reed Army Institute of Research. Although you may withdraw from the study at any time, the samples and data collected up to that time will be used in accordance with the protocol.

Compensation for your participation is provided at each in-person visit. You will not be penalized for stopping your participation early, but we hope you will continue to take part, and we encourage you to remain in contact with the study staff if your situation changes. If you decide to withdraw from the study, please inform the study staff of your decision. We will ask you to attend one final study visit, if you are willing, so that we can make sure that you are safe and that the experimental vaccine is safe. It is important that you let us know how you are doing and if you have any symptoms that might be related to receiving the experimental vaccine. Your well-being is so essential that we ask that you provide us with contact information of a friend or family member just in case we are not able to reach you.

#### What could end my participation in the research?

The study doctor may remove you from the study at any time. This could happen for several reasons, for example, if there is concern about your health, if you do not follow study instructions, or if the sponsor, FDA, or the IRB stop the study. If the study is stopped, the study doctor will inform you. The study could be stopped if there is a safety concern; for example, if one or more participants has a serious reaction that could be considered related to the vaccine, the planned study injections for other participants will be paused to allow the study doctors to look at the data and determine if it is safe to continue. If you miss a study injection for any reason, such as if you are unable to get to the clinic for your study visit, the investigator doesn't think that it is safe for you to receive the injection, or other reasons, you will not be eligible to receive the next study injection. If this happens, we would like you to continue your study visits so that we can make sure you are safe and so that we can assess the safety of the experimental vaccine.

## What if any new information is found out?

During the research, the investigators will tell you of any new findings that might cause you to change your mind about continuing the study. You will be contacted by your preferred method of contact that you wrote down on your intake form, and we will continue our attempts to contact you until we reach you. If we are unable to reach you through your preferred method of contact after 5 attempts, we may attempt contact through your non-preferred methods of contact. It is your responsibility to tell us if your phone number, email, or other contact information changes.

#### Who should I call if I have questions or concerns about this research?

If you have questions about the research at any time or if you have any problems related to the study, you can contact Dr. Brittany Ober-Shepherd by telephone at 260-438-9948 or 301-500-3636, or you can contact the WRAIR CTC study staff at 301-319-9660. An emergency contact card will be provided to you with more numbers to contact at any time.

If you have questions about your rights as a research volunteer in this study, you may contact the WRAIR Human Subjects Protection Branch, 503 Robert Grant Avenue, Silver Spring, MD 20910, phone number 301-319-9940 and email: usarmy.detrick.medcom-wrair.mbx.hspb@health.mil.

If you have any questions or concerns about participating in this study and you are affiliated with the DoD, you can also speak to an ombudsperson who is affiliated with this study. The primary ombudsperson, Ruthie Ratcliffe, can be contacted by telephone at 301-319-3131. If the primary ombudsperson is unavailable, the alternate ombudsperson, Evelina Angov, can be contacted by telephone at 301-319-9614.

## **Study volunteer statement:**

I agree to participate in this study.

I have been asked to take part in the study "A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of Ranging Doses of SARS-CoV-2-Spike-Ferritin-Nanoparticle (SpFN\_1B-06-PL) Vaccine with Army Liposomal Formulation QS21 (ALFQ) for Prevention of COVID-19 in Healthy Adults"

The principal investigator, Dr. Brittany Ober-Shepherd, or her representative, has explained the significance of the testing, the duration of the study, the testing that I will undergo, the methods to be used, and the risks and dangers of participation. I have been informed that by signing this form, I am not giving up any legal rights. I have been given a chance to ask questions about this research study and all questions were answered to my satisfaction. If I have other questions about this research, I can ask Dr. Brittany Ober-Shepherd, by telephone at 260-438-9948 or 301-500-3636 and the WRAIR CTC study staff by telephone at 301-319-9660.

I am signing below to indicate my wish to take part in this study and will follow the requirements of the study as much as possible. I will do my best to follow the recommendations of the study team, and I will report all problems occurring from this study to the study team. It has been explained to me that I can quit this study at any time, and I will not lose any benefits nor will I receive any penalty. The medical care that I could receive as a result of any sickness or injury that may result from being a part of this study have been explained to me and I have been offered a signed copy of this consent form.

| Printed Name of Participant | |
|--------------------------------------|------------|
| Signature of Participant | Date |
| Emergency contact name: | |
| Relation to participant: | |
| Phone number: | |
| Email address: | |
| Printed Name of Person Administering | g Consent |
| Signature of Person Administering C | nsent Date |